CLINICAL TRIAL: NCT00349622
Title: Clinical Trial Ceftriaxone in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Clinical Trial Ceftriaxone in Subjects With ALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Merit E. Cudkowicz, MD, Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U01NS049640-02 (NIH); NINDS (Other: NINDS); U01NS049640-02 (NIH); NINDS CRC (Other: NINDS Clinical Research Collaboration)
Record Dates: First submitted 2006-07-05; First posted 2006-07-07 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: amyotrophic lateral sclerosis; ALS; ceftriaxone; cephalosporin antibiotic; motor neurons
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ceftriaxone (Active Comparator): Two thirds of participants were assigned to 4 grams of ceftriaxone per day. This is a blinded study, so neither participants nor study staff will know which treatment a participant is receiving.
  Ceftriaxone is a cephalosporin antibiotic and was administered intravenously via a central venous catheter twice a day.
  Interventions: Drug: ceftriaxone
- Placebo (Placebo Comparator): One third of participants were assigned to placebo, or an inactive substance. This is a blinded study, so neither participants nor study staff will know which treatment a participant is receiving.
  Pediatric multivitamin solution was used as the placebo in this study and was administered intravenously via a central venous catheter twice a day.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ceftriaxone — Participants will be randomly assigned to receive treatment with ceftriaxone or placebo for at least 12 months. Two thirds of participants will receive ceftriaxone and one third will receive placebo. This is a blinded study, so neither participants nor study staff will know which treatment a participant is receiving.
  Ceftriaxone is approved by the U.S. Food and Drug Administration (FDA) for treating bacterial infections but not for treating ALS. Also, ceftriaxone has not been given to people over a long period of time, such as months or years.
  Arms: Ceftriaxone
Other: placebo — an inactive substance
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of ceftriaxone treatment in amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
It is known that nerve cells called motor neurons die in the brains and spinal cords of people with amyotrophic lateral sclerosis (ALS). However, the cause of this cell death is unknown. Researchers think that increased levels of a chemical called "glutamate" may be related to the cell death. For this reason researchers want to study drugs that decrease glutamate levels near nerves. Ceftriaxone-a semi-synthetic, third generation cephalosporin antibiotic-may increase the level of a protein that decreases glutamate levels near nerves. Studies of ceftriaxone in the laboratory suggest that it may protect motor neurons from injury.

Ceftriaxone is approved by the U.S. Food and Drug Administration (FDA) for treating bacterial infections but not for treating ALS. Also, ceftriaxone has not been given to people over a long period of time, such as months or years. The goals of this study are to evaluate the safety and effectiveness of ceftriaxone as a treatment for ALS, and to determine the safety and effectiveness of long-term use of the drug in people with ALS.

A total of 600 eligible people with ALS will be enrolled in this multi-center research study. Participants will be randomly assigned to receive treatment with ceftriaxone (2/3 of participants) or placebo (1/3 of participants) for at least 12 months.

The study consists of three stages. The first stage, which has completed enrollment, will look at whether ceftriaxone enters the cerebrospinal fluid (the fluid that surrounds the spinal cord, also called CSF) in amounts that are high enough to be of possible benefit. The second stage, which has also completed enrollment, will look at the safety and side effects of the study drug when taken daily for at least 20 weeks. The study is currently enrolling subjects for the third stage, which began in Spring 2009, and will determine whether the study drug prolongs survival and slows decline in function due to ALS.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be people with ALS, at least 18 years of age.
* Participants must be medically able to undergo the study procedures and have a caregiver or other individual who will be available to help with daily study medication administration.
* Participants should live within a reasonable distance of the study site, due to frequent study visits.

Exclusion Criteria:

* Participants cannot be taking any other experimental medications for ALS, or have a history of sensitivity to cephalosporin antibiotics (such as Ancef, Keflex, Ceclor, Ceftin, Lorabid, Suprax, or Fortaz).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2006-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, MSc., Principal Investigator — Associate Professor of Neurology, Harvard Medical School, Massachusetts General Hospital
Locations (58):
- United States (50):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - University of California, Davis, Davis, California
  - University of California, San Francisco- Fresno, Fresno, California
  - Loma Linda University School of Medicine (CA), Loma Linda, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine - MDA ALS Neuromuscular Center, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - ALS Center at Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Northwestern University Medical School, Chicago, Illinois
  - Indiana University (Regenstrief Health Center), Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Saint Mary's Healthcare, Grand Rapids, Michigan
  - Hennepin County Medical Center (Berman Center), Minneapolis, Minnesota
  - St. Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Bryan LGH Medical Center (University of Nebraska), Lincoln, Nebraska
  - UMDNJ- Robert Wood Johnson School of Medicine, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Beth Israel Medical Center (NY), New York, New York
  - Cornell Medical Center, New York, New York
  - Columbia University, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Clinic (Providence Clinic), Portland, Oregon
  - Pennsylvania State University, Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine (Hahnemann Campus), Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Texas Neurology, Dallas, Texas
  - Methodist Neurological Institute, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - Univeristy of Alberta ALS Clinic, Edmonton, Alberta
  - Dalhousie University, Halifax, Nova Scotia
  - London Health Sciences Center, University Campus, London, Ontario
  - University of Toronto, Toronto, Ontario
  - CHUM (Centre Hospitalier de l'Université de Montréal), Notre-Dame Hospital, Montreal, Quebec
  - Montreal Neurological Institute (McGill University), Montreal, Quebec
  - Laval University, Québec, Quebec

REFERENCES:
- [Derived] McDonnell E, Schoenfeld D, Paganoni S, Atassi N. Causal inference methods to study gastric tube use in amyotrophic lateral sclerosis. Neurology. 2017 Oct 3;89(14):1483-1489. doi: 10.1212/WNL.0000000000004534. Epub 2017 Sep 1. PMID 28864675
- [Derived] Cudkowicz ME, Titus S, Kearney M, Yu H, Sherman A, Schoenfeld D, Hayden D, Shui A, Brooks B, Conwit R, Felsenstein D, Greenblatt DJ, Keroack M, Kissel JT, Miller R, Rosenfeld J, Rothstein JD, Simpson E, Tolkoff-Rubin N, Zinman L, Shefner JM; Ceftriaxone Study Investigators. Safety and efficacy of ceftriaxone for amyotrophic lateral sclerosis: a multi-stage, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2014 Nov;13(11):1083-1091. doi: 10.1016/S1474-4422(14)70222-4. Epub 2014 Oct 5. PMID 25297012
- [Derived] Berry JD, Shefner JM, Conwit R, Schoenfeld D, Keroack M, Felsenstein D, Krivickas L, David WS, Vriesendorp F, Pestronk A, Caress JB, Katz J, Simpson E, Rosenfeld J, Pascuzzi R, Glass J, Rezania K, Rothstein JD, Greenblatt DJ, Cudkowicz ME; Northeast ALS Consortium. Design and initial results of a multi-phase randomized trial of ceftriaxone in amyotrophic lateral sclerosis. PLoS One. 2013 Apr 17;8(4):e61177. doi: 10.1371/journal.pone.0061177. Print 2013. PMID 23613806
- See also: Northeast ALS Consortium website — http://www.alsconsortium.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ceftriaxone is approved by the U.S. Food and Drug Administration (FDA) for treating bacterial infections but not for treating ALS. Subjects with ALS were enrolled in 58 institutions across in the US and Canada.
Pre-assignment Details: Participants were randomly assigned to receive treatment with ceftriaxone or placebo for at least 12 months. Two thirds of participants received ceftriaxone and one third received placebo. This is a blinded study, so neither participants nor study staff knew which treatment a participant is receiving.
Period: Overall Study
Arm/Group | Ceftriaxone | Placebo
Started | 340 | 173
Completed | 162 | 77
Not Completed | 178 | 96
Not completed — Death | 168 | 86
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftriaxone | Placebo | Total
Number analyzed (Participants) | 340 | 173 | 513
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age at Screening | 55.6 (10.4) | 54.8 (10.3) | 55.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 72 | 203
  Male | 209 | 101 | 310
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 6 | 23
  Not Hispanic or Latino | 320 | 165 | 485
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 3 | 11
  White | 320 | 163 | 483
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 293 | 151 | 444
  Canada | 47 | 22 | 69
ALS Family History [Number; unit: participants] — Subjects were asked at screening whether or not they have a familial history of ALS.
  participants
    Familial History of ALS | 26 | 8 | 34
    No Known Familial History of ALS | 307 | 161 | 468
    Unknown | 7 | 4 | 11
Site of Onset [Number; unit: participants] — Indicates region of first symptoms
  participants
    Limb | 257 | 137 | 394
    Bulbar | 75 | 35 | 110
    Both | 8 | 1 | 9
Riluzole Use [Number; unit: participants] — At the screening visit, subjects were asked whether or not they were taking a continuous dose of riluzole.
  participants
    On Riluzole | 249 | 128 | 377
    Not on Riluzole | 91 | 45 | 136
Vital Capacity Percent Predicted [Mean (Standard Deviation); unit: percent predicted based on age and heigh] — The vital capacity (lung capacity) for each subject was measured at screening.
  percent predicted based on age and heigh | 87.9 (16.6) | 91.1 (18.4) | 89.0 (17.3)
Time to Screening [Mean (Standard Deviation); unit: years]
  Years from Symptom Onset to Screening | 1.49 (0.68) | 1.50 (0.67) | 1.49 (0.68)
  Years from Diagnosis to Screening | 0.56 (0.49) | 0.58 (0.49) | 0.57 (0.49)
  Years from Symptom Onset to Diagnosis | 0.93 (0.55) | 0.92 (0.58) | 0.92 (0.56)

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Survival is presented as median day of survival for each group. Survival is defined as time to death, tracheostomy or the initiation of permanent assisted ventilation (PAV).
Time Frame: From date of randomization until date of death, tracheostomy, or the initiation of permanent assisted ventilation (PAV). This was assessed at time of each participant's drug discontinuation and every 2 months thereafter for the life of the study (6 yrs)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 340 | 173
days | 664 [614 to 794] | 581 [521 to 672]

2. Primary Outcome: Change From Baseline in ALS Functional Rating Scale, Revised (ALSFRS-R) at One Year
Description: Amyotrophic Lateral Sclerosis Functional Rating Scale, Revised (ALSFRS-R) is a quickly administered (five minute) ordinal rating scale used to determine patients' assessment of their capability and independence in 12 functional activities/questions. The 12 functional activities/questions are rated on a scale of 0 to 4 for a total scoring range of 0-48, with 48 representing optimal function. All 12 activities are relevant in ALS.
  This outcome measure calculation is based on measurements every 8 weeks from the Baseline Visit up until one year.
Time Frame: Every 8 weeks for one year
Measure: Mean (Standard Error); unit: units on a scale per 8 weeks
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 340 | 173
units on a scale per 8 weeks | -1.1311 (0.04395) | -1.2208 (0.06177)

3. Secondary Outcome: Change in % Vital Capacity From Screening to One Year
Description: Vital Capacity is measured as the percent predicted per subject based on age, gender, and height, and is performed as a Slow Vital Capacity.
  This outcome measure calculation is based on measurements every 12 weeks from the Baseline Visit up until one year.
Time Frame: Every 12 weeks for one Year
Measure: Mean (Standard Error); unit: percent change in VC per 12 weeks
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 340 | 173
percent change in VC per 12 weeks | -2.772 (0.1417) | -3.0826 (0.1970)

4. Secondary Outcome: Change From Baseline in Evaluation of Multiple Upper Extremity Muscles Using Hand Held Dynamometry at One Year
Description: Hand-held Dynamometry (HHD) is used to evaluate muscle strength. Six proximal muscle groups were examined bilaterally in both upper and lower extremities (shoulder flexion, elbow flexion, elbow extension, hip flexion, knee flexion, and knee extension). In addition, wrist extension, first dorsal interosseous contraction and ankle dorsiflexion were measured bilaterally.
  HHD analysis was performed using Percent Change from Baseline. Each subject's baseline strength value for each muscle group is considered 100%. During successive visits strength for each muscle group was measured using HHD and was calculated as a percentage of the initial baseline value recorded. Upper extremity and lower extremity values were calculated as the sum of all tests for that extremity to create one megascore for upper and one megascore for lower extremity muscles.
  This outcome measure calculation is based on measurements every 12 weeks from the Baseline Visit up until one year.
Time Frame: Every 12 weeks for one Year
Measure: Mean (Standard Error); unit: Percent change per 12 weeks
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 340 | 173
Percent change per 12 weeks | -5.2735 (0.2178) | -5.5526 (0.3040)

5. Secondary Outcome: Change From Baseline in the ALS-Specific Quality of Life Scale (ALSQOL) at One Year
Description: The ALS-Specific Quality of Life Scale (ALSQOL). was developed, tested, and validated in subjects with ALS, and is not a health-related quality of life scale. The scale consists of 59 questions that ask about severity of the symptoms of ALS, mood and affect, intimacy, and social issues. Each question for the ALSQOL is scored from 0-10. With 59 questions, total score ranges from 0-590 with scores simply added, with 590 representing highest quality of life. However since 10 is maximally weighted towards negative values on some questions and positive values on others, the following questions must have results transposed (Simply reverse the scale, for instance 10=0 and 0=10) prior to analysis: 1-10, 11, 16, 19, 24, 26, 28, 32, 35, 36, 38, and 41. Optional items are 50, 53, 56, and 59. These questions are not included on any scale or in any quantitative analyses.
  This outcome measure calculation is based on measurements every 12 weeks from the Baseline Visit up until one year.
Time Frame: Every 12 weeks for one Year
Measure: Mean (Standard Error); unit: units on a scale per 12 weeks
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 340 | 173
units on a scale per 12 weeks | -3.5084 (0.3297) | -3.4401 (0.4629)

6. Secondary Outcome: Change From Baseline in Evaluation of Multiple Lower Extremity Muscles Using Hand Held Dynamometry at One Year
Description: as for outcome 4
Time Frame: Every 12 weeks for one Year
Measure: Mean (Standard Error); unit: Percent change per 12 weeks
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 340 | 173
Percent change per 12 weeks | -4.1530 (0.2591) | -4.4807 (0.3625)

ADVERSE EVENTS:
Time Frame: Adverse Events were systematically assessed by study investigators at each study visit from the screening visit until 30 days after permanent study drug discontinuation. The total amount of time per subject varies by length of subject participation.
Description: Adverse Events were systematically assessed by study investigators at each study visit from the screening visit until 30 days after permanent study drug discontinuation.
Arm/Group | Ceftriaxone | Placebo
Serious Adverse Events (participants affected / at risk) | 276/340 | 125/173
Other Adverse Events (participants affected / at risk) | 331/340 | 153/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftriaxone (N=340) | Placebo (N=173)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 74 (79) | 34 (35)
Cholelithiasis (Hepatobiliary disorders) | 28 (30) | 0 (0)
Infections with unknown ANC: Lung (pneumonia) (Infections and infestations) | 13 (17) | 12 (14)
Thrombosis/thrombus/embolism (Vascular disorders) | 20 (20) | 4 (4)
Line Infection (Infections and infestations) | 3 (4) | 9 (11) — "Line Infection" was added to the trial database as an adverse event potentially related to the central venous catheter that all subjects received as part of the study.
Renal/Genitourinary - Other (Renal and urinary disorders) | 10 (10) | 1 (1)
PEG Placement (outpatient) (Surgical and medical procedures) | 4 (4) | 5 (6) — PEG (Percutaneous Endoscopic Gastrostomy) Placement was added as an adverse event term during STAGES 1 and 2 of this study. PEG tube placements are common for people with ALS. In STAGE 3 of the study, these events were coded as Dysphagia.
Aspiration (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Death not associated with CTCAE Term: Disease Progression NOS (General disorders) | 4 (4) | 4 (4)
Cardiac ischemia/infarction (Cardiac disorders) | 6 (8) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Infection with normal ANC or grade 1 or 2 neutrophils: Lung (pneumonia) (Infections and infestations) | 4 (4) | 2 (2)
Catheter Exit Site Infection (Infections and infestations) | 2 (2) | 3 (3) — "Catheter Exit Site Infection" was added to the trial database as an adverse event potentially related to the central venous catheter that all subjects received as part of the study.
Cholecystitis (Hepatobiliary disorders) | 5 (5) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4 (4) | 0 (0)
Death not associated with CTCAE term: Death NOS (General disorders) | 3 (3) | 1 (1)
Fever (in the absense of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 2 (2) | 2 (2)
Infection with normal ANC or grade 1 or 2 neutrophils: Blood (Infections and infestations) | 1 (1) | 3 (3)
Infections with unknown ANC: Blood (Infections and infestations) | 1 (1) | 3 (3)
Pain: Abdomen NOS (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Colitis infectious (Clostridium difficile) (Infections and infestations) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal - Other (Gastrointestinal disorders) | 0 (0) | 3 (3)
Infection with unknown ANC: Urinary tract NOS (Infections and infestations) | 0 (0) | 3 (3)
Joint-function (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 1 (1)
Death not associated with CTCAE Term: Sudden Death (General disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Line break/tear (General disorders) | 2 (2) | 0 (0) — "Line break/tear" was added to the trial database as an adverse event potentially related to the central venous catheter that all subjects received as part of the study.
Line Displacement (General disorders) | 1 (1) | 1 (1) — "Line Displacement" was added to the trial database as an adverse event potentially related to the central venous catheter that all subjects received as part of the study.
Mood alteration: Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neurology - Other (Nervous system disorders) | 1 (1) | 1 (1)
Obstruction/stenosis of airway: Larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Biliary Sludge (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cardiac/Arrhythmia Other (Cardiac disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
FEV (1) (Investigations) | 0 (0) | 1 (1)
Febrile neutropenia (fever of unknown origin w/out clinically/microbiologically documented infection (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn/Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemmorhage, CNS (Nervous system disorders) | 0 (0) | 1 (1)
Hemmorhage, GI: Lower GI NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemmorhage, GI: Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemmorhage, pulmonary/Upper Respiratory: Stoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hemorrhage/bleeding associated with surgery, intraoperative or postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatobiliary - Other (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia: Lung (Infections and infestations) | 0 (0) | 1 (1)
Infection - Other (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or grade 1 or 2 neutrophils: Bronchus (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or grade 1 or 2 neutrophils: Vagina (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC: Abdomen NOS (Infections and infestations) | 1 (2) | 0 (0)
Infection with unknown ANC: Catheter-related (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC: Foreign body (e.g. graft, implant, prosthesis, stent) (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC: Soft tissue NOS (Infections and infestations) | 0 (0) | 1 (1)
Leak (including anastomotic), GI: Stomach (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Line Thrombosis (General disorders) | 1 (1) | 0 (0) — "Line Thrombosis" was added to the trial database as an adverse event potentially related to the central venous catheter that all subjects received as part of the study.
Metabolic/Laboratory - Other (Investigations) | 1 (1) | 0 (0)
Mood alteration: Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Mood alteration: Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1) | 0 (0)
Obstruction, GI: Ileum (Gastrointestinal disorders) | 1 (2) | 0 (0)
Obstruction, GI: Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction/stenosis of airway: Trachea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain: chest wall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain: Chest/thorax NOS (General disorders) | 1 (1) | 0 (0)
Pain: Head/headache (Nervous system disorders) | 1 (1) | 0 (0)
Pain: Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Potassium, serum-low (hypokalemia) (Investigations) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Sexual/Reproductive Function - Other (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Stricture/stenosis (including anastomotic), GU: Ureter (Renal and urinary disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmias: Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 1 (1)
Urinary retention (including nerogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia: Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 7 (7) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftriaxone (N=340) | Placebo (N=173)
Diarrhea (Gastrointestinal disorders) | 152 (220) | 41 (51)
Cholelithiasis (Hepatobiliary disorders) | 158 (193) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 32 (38) | 24 (26)
Neurology - Other (Nervous system disorders) | 97 (183) | 52 (92)
Catheter Exit Site Reaction (General disorders) | 98 (143) | 45 (69) — "Catheter Exit Site Reaction" was added to the trial database as an adverse event potentially related to the central venous catheter that all subjects received as part of the study.
Rash/desquamation (Skin and subcutaneous tissue disorders) | 92 (122) | 29 (36)
Biliary Sludge (Hepatobiliary disorders) | 100 (110) | 12 (12)
Constipation (Gastrointestinal disorders) | 66 (76) | 30 (34)
Pain: Abdomen NOS (General disorders) | 75 (114) | 16 (17)
Nausea (Gastrointestinal disorders) | 64 (115) | 28 (39)
Pain: head/headache (Nervous system disorders) | 53 (79) | 32 (37)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 57 (78) | 21 (25)
Edema: Limb (General disorders) | 54 (68) | 22 (25)
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 46 (61) | 26 (30)
Pain: Back (Musculoskeletal and connective tissue disorders) | 53 (59) | 17 (22)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 46 (57) | 20 (25)
Pain: Joint (Musculoskeletal and connective tissue disorders) | 47 (62) | 19 (24)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 41 (44) | 24 (26)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 45 (57) | 17 (24)
Insomnia (Psychiatric disorders) | 40 (42) | 19 (19)
Dysphagia, (difficult swallowing) (Gastrointestinal disorders) | 35 (38) | 17 (17)
Infection - Other (Infections and infestations) | 42 (64) | 15 (18)
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-upper (Musculoskeletal and connective tissue disorders) | 39 (48) | 19 (22)
Renal/Genitourinary - Other (Renal and urinary disorders) | 37 (57) | 13 (20)
Mood alteration: Depression (Psychiatric disorders) | 33 (33) | 21 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 41 (48) | 12 (15)
Gastrointestinal - Other (Gastrointestinal disorders) | 36 (41) | 12 (16)
Mood alteration: Anxiety (Psychiatric disorders) | 34 (38) | 14 (14)
Pain: Neck (General disorders) | 34 (37) | 15 (17)
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 38 (53) | 10 (12)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 33 (41) | 14 (14)
Drooling (Nervous system disorders) | 30 (30) | 16 (16)
Infection with normal ANC or grade 1 or 2 neutrophils: Urinary Tract NOS (Infections and infestations) | 25 (29) | 17 (24)
Dizziness (Nervous system disorders) | 25 (32) | 15 (18)
Fever (absence of neutropenia, where neutropenia is AGC <1.0x10e9/L) (General disorders) | 27 (28) | 12 (15)
ALT SGPT (serum glutamic pyruvic transaminase) (Investigations) | 32 (42) | 5 (6)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 14 (16)
Pain: chest wall (Musculoskeletal and connective tissue disorders) | 25 (29) | 12 (17)
Heartburn/Dyspepsia (Gastrointestinal disorders) | 24 (26) | 12 (14)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration of voice, laryngitis) (Nervous system disorders) | 25 (27) | 11 (11)
Muscle weakness, generalized of specific area (not due to neuropathy): Whole body/generalized (Musculoskeletal and connective tissue disorders) | 27 (29) | 8 (9)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 24 (44) | 10 (15)
Fracture (Injury, poisoning and procedural complications) | 24 (29) | 10 (11)
Vomiting (Gastrointestinal disorders) | 24 (33) | 10 (13)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 30 (41) | 2 (2)
Metabolic/Laboratory (Investigations) | 18 (22) | 13 (20)
Urinary frquency/urgency (Renal and urinary disorders) | 20 (21) | 11 (13)
Line break/tear (General disorders) | 19 (21) | 11 (12) — "Line break/tear" was added to the trial database as an adverse event potentially related to the central venous catheter that all subjects received as part of the study.
Pain - Other (General disorders) | 18 (26) | 12 (13)
Infection with unknown ANC: Upper airway NOS (Infections and infestations) | 20 (34) | 9 (10)
Infection with unkown ANC: Urinary tract NOS (Infections and infestations) | 17 (18) | 11 (15)
AST SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 23 (27) | 4 (5)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 19 (25) | 7 (7)
Weight loss (Investigations) | 15 (16) | 11 (11)
Hepatobiliary - Other (Hepatobiliary disorders) | 20 (25) | 5 (6)
Hypertension (Vascular disorders) | 16 (22) | 9 (9)
Lymphopenia (Blood and lymphatic system disorders) | 20 (24) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No